CLINICAL TRIAL: NCT07191080
Title: Application of Respiratory Specimens mNGS and tNGS in Aetiological Diagnosis
Brief Title: Next-generation Sequencing Technology in the Clinical Application of Respiratory Specimens
Status: Enrolling by invitation | Type: Observational
Sponsor: Bin Zhang (Other)
Responsible Party: Sponsor-Investigator, Bin Zhang, Chief physician, Affiliated Hospital of Nantong University
Organization: Affiliated Hospital of Nantong University (Other)
Other Study IDs: MSZ2023197
Record Dates: First submitted 2025-07-21; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Lung Infection
Keywords: mNGS; tNGS; Severe lung infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obtain the performance parameters and clinical consistency of mNGS and tNGS technologies in the pathogen diagnosis of lower respiratory tract specimens from patients with severe pulmonary infections, to provide a reference basis for the application value and true performance of these technologies in the pathogen diagnosis of patients with severe pulmonary infections.

DETAILED DESCRIPTION:
Compared with pathogenic mNGS detection of lower respiratory tract airway secretion specimens, pathogenic tNGS detection can further shorten the detection time.It can more accurately analyze the pathogen composition of the patient's lower respiratory tract infectious diseases and identify the diagnostic results of the pathogen of lower respiratory tract infections.It also has a very high accuracy in identifying atypical special pathogens such as fastidious bacteria, fungi and viruses.

This study plans to enroll patients with severe pulmonary infection admitted to the Affiliated Hospital of Nantong University, and collect samples of alveolar lavage fluid or sputum specimens collected by the airway specification from the patients will be sent for testing of mNGS and tNGS, the results obtained from different methodological tests will be compared and analyzed, and the clinical data of patients (including basic information of patients (including gender, age, height, weight, past medical history, etc.), traditional pathogen testing, G/GM experiments, blood routine, PCT, CRP, CD4 lymphocytes, IFN, IL-6, IL-2 and serum antigen detection, clinical antimicrobial drug use, imaging examination, etc.) will be collected through the electronic medical record system. The test results will be analyzed and compared with the clinical condition of the patients, and finally the detection performance of mNGS and tNGS will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of the informed consent form.
2. Common respiratory infections: traditional methods cannot clearly identify and the patient's condition is prolonged without improvement; Patients with a high suspicion of viral pneumonia: such as acute onset during a season of high viral incidence, normal or low blood leukocyte counts, rapid disease progression, negative results for respiratory viral multiplex PCR testing and cultures; Immunocompromised patients: experiencing respiratory infections or severe illness.
3. Sufficient samples can be obtained.
4. Patients with complete clinical data.

Exclusion Criteria:

1. Refusal to sign informed consent.
2. Testing has clearly excluded infection.
3. Received antibiotic treatment within three days prior to testing without stopping the medication for more than 12 hours.
4. Sample quality is not up to standard.
5. Unable to obtain sufficient sample.
6. No complete drug usage history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe pulmonary infections from the Affiliated Hospital of Nantong University.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison the results of the microbial detection rates of mNGS and tNGS、the number of strains detected and the type number of species detected | The time from the enrollment test to the result ,usually within 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No